CLINICAL TRIAL: NCT05412758
Title: Augmented Response of Volatile Biomarkers in Assessment of Oesophagogastric Cancer
Brief Title: Augmented Response of Volatile Biomarkers in Assessment of Oesophagogastric Cancer (AROMA 1 / BIORESOURCE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); University Hospital Plymouth NHS Trust (Other); Royal Surrey County Hospital NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); Barking, Havering and Redbridge University Hospitals NHS Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); University College London Hospitals (Other); Cardiff and Vale University Health Board (Other Government); NHS Lothian (Other Government); NHS Tayside (Other Government); York Teaching Hospitals NHS Foundation Trust (Other); The Harley Street Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21HH7100
Record Dates: First submitted 2022-04-01; First posted 2022-06-09 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Volatile Organic Compounds; Microbiome; Microbioata; Breath Analysis; Oesophageal Cancer; Gastric Cancer; Volatalomics; Metabonomics/Lipidomics; Microbiome Analysis; Transcriptomics
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: There are two arms to this study; AROMA 1 and BIORESOURCE. It is the AROMA 1 arm of the study that involves an intervention. A total of 648 patients will be recruited for development of an augmented breath test to detect oesophageal and gastric cancer at early stages of disease. Three groups, each containing 216 patients, will be recruited: (i) oesophageal cancer (ii) gastric cancer and (iii) control/normal patients with upper gastrointestinal symptoms. After the first baseline breath sample at 0 minutes is collected, subjects will then be asked to consume a standard nutrient drink. Further breath samples will be collected at 15 minutes after consumption of the drink.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oesophageal/GOJ cancer (Experimental): AROMA 1: 216 treatment naive patients with oesophageal/GOJ cancer will be recruited to undertake an augmented breath test.
  BIORESOURCE: 110 treatment naive patients with oesophageal/GOJ cancer will be recruited for biosample collection at the time of their staging laparoscopy procedure.
  Interventions: Dietary Supplement: Oral Stimulant Drink
- Gastric cancer (Experimental): AROMA 1: 216 treatment naive patients with gastric cancer will be recruited to undertake an augmented breath test.
  BIORESOURCE: 75 treatment naive patients with gastric cancer will be recruited for biosample collection at the time of their staging laparoscopy procedure.
  Interventions: Dietary Supplement: Oral Stimulant Drink
- Control/ normal patients with upper gastrointestinal symptoms (Experimental): AROMA 1: 216 control subjects will be recruited to undertake an augmented breath test.
  BIORESOURCE: 150 control subjects will be recruited for biosample collection at the time of their routine endoscopy procedure.
  Interventions: Dietary Supplement: Oral Stimulant Drink

INTERVENTIONS:
Dietary Supplement: Oral Stimulant Drink — For the AROMA 1 study patients will be requested to consume a nutrient drink (approximately 200 ml) that includes natural ingredients found within a typical human diet. Following consumption of the drink, serial breath tests will be performed to determine varying levels of VOC production in breath
  Other Names: Oral Nutrient Drink

SUMMARY:
Cancer of the stomach and oesophagus is among the world's top five cancers. Survival rates are very poor as the disease presents late and early symptoms are non-specific. The study team has developed a non-invasive test for cancers of the stomach and oesophagus based on the detection of volatile organic compounds in exhaled breath. These compounds are known to be produced by both cancers as well as cancer associated bacteria within the gut.

The proposed innovation is to improve the accuracy of this test by investigating whether simple metabolic substrates can increase the production of these volatile organic compounds by both the tumour and its associated bacteria.

DETAILED DESCRIPTION:
AROMA 1: A total of 648 patients will be recruited for development of an augmented breath test to detect oesophageal and gastric cancer at early stages of disease. Three groups, each containing 216 patients, will be recruited: (i) oesophageal cancer (ii) gastric cancer and (iii) control/normal patients with upper gastrointestinal symptoms. After a baseline breath sample is collected, subjects will then be asked to consume a standard nutrient drink. Further breath samples will be collected at 0 and 15 minutes after consumption of the drink.

Breath samples will be stored on thermal desportion tubes before being transfered to a central laboratory for analysis. Breath samples will be analysed in accordance with existing quality-controlled processes. A combined approach of chromatographic- and real time- mass spectrometric techniques will be applied for VOC profiling.

BIORESOURCE: Samples from 335 patients will be collected in order to establish a biobank for multi-omic analyses. Three groups, each containing 75 patients, will be recruited: (i) oesophageal adenocarcinoma; (ii) gastric adenocarcinoma and (iii) oesophageal controls - benign conditions/normal gastrointestinal tract with upper gastrointestinal symptoms (iv) gastric controls - benign conditions/normal gastrointestinal tract with upper gastrointestinal symptoms. The following biosamples will be collected: breath, urine, saliva, blood, tissue and gastric contents. Collected samples will be utilised in a wide range of studies to investigate the mechanisms of VOC production in cancer. The following analyses will be performed: volatalomics, metabonomics/lipidomics, microbiome analysis, transcriptomics and cell culture experiments.

ELIGIBILITY:
AROMA 1 Inclusion Criteria:

1. Aged 18-90years
2. Oesophageal/gastric cancer cohort: participants with biopsy proven adenocarcinoma who are treatment naïve
3. Control cohort: participants with normal or benign upper gastrointestinal disease determined on: • Endoscopy within 1 year • Planned endoscopy

AROMA 1 Exclusion criteria:

Patients with the following characteristics will not be eligible for inclusion in this study:

1. Oesophageal squamous cell carcinoma
2. Previous oesophageal and gastric resection
3. Received neoadjuvant chemotherapy for oesophageal or gastric cancer
4. History of another cancer within three years
5. Any form of oesophageal dysplasia (control cohort only)
6. Previously diagnosed with Barrett's oesophagus (control cohort only)
7. Active infection, on immunosuppressive medications or antibiotic therapy within the last 8 weeks
8. Participants with co-morbidities preventing breath collection
9. Allergies to any of the constituents of the nutrient drink including glucose, glycerol, iron sulphate, Maltodextrin (Corn, Potato), Xanthan Gum, Potassium Chloride, tyrosine, phenylalanine, and glutamic acid
10. Unable or unwilling to provide informed written consent
11. Pregnant participants

BIORESOURCE inclusion criteria:

1. Aged 18- 90years
2. Oesophageal/gastric cancer cohort: participants with biopsy proven adenocarcinoma who are treatment naïve
3. Oesophageal/gastric control cohort: participants with normal or benign upper gastrointestinal disease determined on: • Planned endoscopy

BIORESOURCE exclusion criteria:

1. Oesophageal squamous cell carcinoma
2. Previous oesophageal and gastric resection
3. Received neoadjuvant chemotherapy for oesophageal or gastric cancer
4. History of another cancer within five years
5. Any form of oesophageal dysplasia (oesophageal/gastric control cohorts only)
6. Previously diagnosed with Barrett's oesophagus (oesophageal/gastric control cohorts only)
7. Active infection, on immunosuppressive medications or antibiotic therapy within the last 8 weeks
8. Participants with co-morbidities preventing breath collection
9. Unable or unwilling to provide informed written consent
10. Pregnant participants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of an oral nutrient drink to stimulate the production of volatile organic compounds detected in the breath. | 18 months
  Efficacy of the oral stimulant drink will be measured by comparing the relative abundance of certain volatile organic compounds (measured in ppt) detected in the breath. Breath analysis will be performed with the help of Gas Chromatography- Mass Spectrometry (GC-MS)

SECONDARY OUTCOMES:
Volatile metabolites present in breath of subjects with oesophagogastric cancer and controls | 18 months
  GC-MS will be used to determine the presence of certain cancer associated volatile organic compounds in breath
Volatile metabolites present in headspace of the urine of subjects with oesophagogastric cancer and controls | 18 months
  Headspace sampling techniques will be used for headspace collection from urine samples. GC-MS will be used to determine the presence of certain cancer associated volatile organic compounds within the headspace of urine.
Determination of bacterial species and cancer associated volatile compound production from saliva samples of subjects with oesophagogastric cancer. | 18 months
  Bacterial species will be determined using sequencing techniques such as 16s or whole genome sequencing. Bacteria within the saliva samples will be cultured and species isolated. Once isolated, cancer associated species will be re-cultured within a controlled environment. Headspace and media sampling will be performed to determine the volatile metabolites present using GC-MS and LC-MS techniques
Determination of bacterial species and cancer associated volatile compound production from tissue samples of subjects with oesophagogastric cancer | 18 months
  Bacterial species will be determined using sequencing techniques such as 16s or whole genome sequencing. Tissue and bacteria from biopsies will be separated. Bacteria derived from tissue samples will be cultured and species isolated. Once isolated, cancer associated species will be re-cultured within a controlled environment. Headspace and media sampling will be performed to determine the volatile metabolites present using GC-MS and LC-MS techniques
Determination of bacterial species and cancer associated volatile compound production from gastric contents of subjects with oesophagogastric cancer | 18 months
  Bacterial species will be determined using sequencing techniques such as 16s or whole genome sequencing. Bacteria from gastric content samples will be separated. Bacteria derived from gastric juices will be cultured and species isolated. Once isolated, cancer associated species will be re-cultured within a controlled environment. Headspace and media sampling will be performed to determine the volatile metabolites present using GC-MS and LC-MS techniques

CONTACTS AND LOCATIONS:
Overall Officials: George Hanna, PhD, FRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No